CLINICAL TRIAL: NCT07096050
Title: Post Marketing Clinical Follow up Study to Evaluate the Performance and Safety of HyaleXo for Pain Relief in Patients Suffering From Osteoarthritis or Degenerative Joint Diseases
Brief Title: Post Marketing Clinical Follow up Study of HyaleXo
Acronym: PMCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Collaborators: TigerMed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YYDATP-PMCF-RO
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients that meet inclusion/exclusion criteria. (Other): Patients that meet inclusion/exclusion criteria.
  Interventions: Other: HyaleXo

INTERVENTIONS:
Other: HyaleXo — Treatment of HyaleXo 3 times

SUMMARY:
Hyaluronic acid is a polysaccharide naturally present in several human tissues such as cartilage. It is the major constituent of synovial fluid and provides its viscosity and elasticity. In traumatic and degenerative joint diseases, the amount of hyaluronic acid is reduced. The consequent loss of viscosity by the synovial fluid may be the cause of painful symptoms. HyaleXo action, according to its composition (sodium hyaluronate of very high molecular weight), may restore the viscoelastic properties of synovial fluid, attenuate pain and improve the mobility of the joint. These characteristics allow HyaleXo to be used for the symptomatic relief of pain in patients suffering from osteoarthritis (OA) or degenerative joint diseases causing an alteration of the functionality of the synovial fluid.

The patient will be treated with HyaleXo as reported in the Instruction for use (IFU) of the device: via injection once a week for 3 weeks using standard technique. The patient pain management strategy should be according to the standard clinical practices and remains at the discretion of the investigator.

The Research Question of the present study is the following: in a population of men and women suffering from painful knee osteoarthritis or degenerative joint disease will very high molecular weight fraction of sodium Hyaluronate (HyaleXo) significantly decrease and / or relieve the pain after 1,6,12 weeks and 6 months of the third injection?

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years old (inclusive ≥ 18 years).
2. Men or women.
3. Patients suffering from painful chronic idiopathic symptomatic degenerative joint diseases (clinical evidence) OR knee osteoarthritis (as defined by the American College of Rheumatology (ACR) criteria); for patients with OA at both knees, only the most painful one will be included in the study.
4. VAS knee pain ≥ 40 mm at screening and 30 days before.
5. Patients willing and able to comply with study terms.
6. Patients willing to discontinue all other OA treatments

Exclusion Criteria:

1. Patients that are unable or unwilling to provide informed consent, and/or patients participating in a concurrent clinical trial and/or patients who have participated in a similar clinical trial within the last days.
2. Patients with known hypersensitivity to any components of investigational product.
3. Patients who are pregnant or breastfeeding. Patients with infected or severely inflamed joints.
4. Patients with skin diseases or infections in the area of the injection site.
5. Patients with hepatic failure or history thereof.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Functional assessment of HyaleXo by KOOS | 12 weeks
  Functional assessment of HyaleXo by KOOS (Knee Injury and Osteoarthritis Outcome score) for Pain subscale at 12 weeks after the last administration of the investigational product, compared to the baseline.

SECONDARY OUTCOMES:
Functional assessment of HyaleXo by KOOS | 1,6,12 weeks and 6 months
  Functional Assessment of HyaleXo by KOOS for other Symptoms, Activity of Daily Living (ADL), Sport and Recreation (Sport/Rec) function and knee related Quality of life (QoL) at 1, 6, 12 weeks and 6 months after the last administration of the investigational product, compared to baseline
Functional assessment of HyaleXo by KOOS | 1,6 weeks and 6 months
  Functional Assessment of HyaleXo by KOOS for Pain subscale at 1, 6 weeks and 6 months after the last administration of the investigational product, compared to baseline
Visual Analgoue Sclae | 1,6,12 weeks and 6 months
  • Changes in the weight-bearing pain using a Visual Analogue Scale (100 mm - VAS) at 1, 6, 12 weeks and 6 months after the last administration, compared to the baseline.
Visual Analgoue Sclae | 1,6,12 weeks and 6 months
  • Changes in the rest pain (100 mm - VAS) at 1, 6, 12 weeks and 6 months after the last administration, compared to the baseline.
Visual Analgoue Sclae | 1,6,12 weeks and 6 months
  • Changes in the motion pain (pain after 15 m walk) (100 mm - VAS) at 1, 6, 12 weeks and 6 months after the last administration, compared to the baseline.
Patient Global Pain Assessment | 1,6,12 weeks and 6 months
  • Patient Global Pain Assessment (100 mm - VAS) at 1, 6, 12 weeks and 6 months after the last administration, compared to the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Echipa Medical 33, Timișoara, Romania

IPD SHARING:
Plan to Share IPD: No